CLINICAL TRIAL: NCT03788044
Title: Effect of Targeted Education for Atrial Fibrillation Patients (Application Substudy)
Acronym: AF-EduApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Bristol-Myers Squibb (Industry); Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Hein Heidbuchel, Professor Doctor, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF-EduApp / EC 18/12/171; CV185-696 (Other Grant/Funding Number: ERISTA (European Thrombosis Investigator Initiated Research Program) grant supported by BMS/Pfizer)
Record Dates: First submitted 2018-12-05; First posted 2018-12-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation and Flutter
Keywords: Education; Application; Adherence
MeSH Terms: conditions — Atrial Fibrillation | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: AF patients will be divided in four groups (AF-EduCare study and AF-EduApp substudy): one group will have application-based education (AF-EduApp substudy), the second group will have in-person education (AF-EduCare study), the third group will have online education (AF-EduCare study) and the fourth group will receive standard AF care (AF-EduCare study and not eligible for AF-EduApp substudy). NOAC adherence will be compared between these groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Application-driven education (AF-EduApp substudy) (Experimental): Education will be given via a newly developed application. Medication adherence (oral anticoagulation) will be measured using a special bottle cap that fits on a medication bottle. The patients in this group will receive feedback (notification and/or alarm) during the entire study period via this application when these patients have to take their medication.
  Interventions: Other: Education
- In-person education (AF-EduCare study) (Experimental): Education will be given on regular basis via predefined consultation visits. Medication adherence (oral anticoagulation) will also be measured using a special bottle cap that fits on a medication bottle. If adherence is low, the patient will get additional feedback when he does not take this medication as prescribed.
  Interventions: Other: Education
- Online education (AF-EduCare study) (Experimental): Education will be given on regular basis via a special designed online platform. Medication adherence (oral anticoagulation) will also be measured using a special bottle cap that fits on a medication bottle. If adherence is low, the patient will get additional feedback when he does not take this medication as prescribed.
  Interventions: Other: Education
- Standard care (AF-EduCare study and AF-EduAppsub study) (No Intervention): This group of AF patients will serve as a control group and no extra focused educational reinforcements will be provided beyond standard care (i.e. information of the treating physician and a brochure).

INTERVENTIONS:
Other: Education — Education + Medication adherence monitoring + Feedback when low adherence
  Arms: Application-driven education (AF-EduApp substudy); In-person education (AF-EduCare study); Online education (AF-EduCare study)

SUMMARY:
The aim of this study is to evaluate a new and innovative educational application based on targeted education on the adherence level for NOACs (non-vitamin K antagonist oral anticoagulants) in AF patients, compared with standard care, online targeted education and in-person targeted education.

Several other parameters (knowledge level, quality of life, symptom burden, self-care capabilities, evaluation of educational efforts) will be studied. If resources allow, cardiovascular outcomes, cost-effectiveness and cost-utility will also be investigated.

DETAILED DESCRIPTION:
This substudy is part of the AF-EduCare study (NCT03707873): an extra study arm will be added to the main trial in which eligible AF patients (= in possession of a smartphone and capable working with their smartphone) will test this new educational application. Not eligible patients randomized to this group, will receive standard care.

This extra study arm will additionally include an anticipated 221 patients (eligible plus not eligible patients).

[An anticipated total of 1259 AF patients will be included for the AF-EduCare study (1038 AF patients) plus the AF-EduApp substudy (221 AF patients).]

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients in whom AF or atrial flutter is diagnosed with an electrocardiogram (12-lead, holter,...).
3. Patients who are capable to sign the informed consent.

Exclusion Criteria:

1. Not able to speak and read Dutch.
2. Cognitive impaired (e.g. severe dementia).
3. Life expectancy is estimated to be less than 1 year.
4. Ongoing participation in another clinical trial.
5. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Patients' adherence to medication (oral anticoagulation), measured by the Medication Events Monitoring System (MEMS). | Monitored between 0-12 months and 12-15 months if resources allow.

SECONDARY OUTCOMES:
Patients' knowledge level, assessed by the Jessa Atrial fibrillation Knowledge Questionnaire (JAKQ) | at baseline,1 month,3-,6-,12 months in the application group.(+18-and if applicable at 24-,30-,36 months/at the end of the study in the other intervention groups).In the standard care groups at 12 or 18 months (if applicable at the end of the study).
  This questionnaire includes 16 knowledge questions: 8 about atrial fibrillation, 5 about oral anticoagulation medication and 3 about vitamine K antagonists or non-vitamin K antagonist oral anticoagulants. A total score between 0% and 100% will be generated in which 100% is the best possible score (all questions are answered correctly).
Patients' quality of life, assessed by the EQ-5D-3L questionnaire and the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire. | at baseline, 3- and 12 months in the application group.(+18-and if applicable at 36 months/at the end of the study in the other intervention groups.) In the standard care groups at baseline and 12 or 18 months (and if applicable at the end of the study).
  The EQ-5D-3L descriptive system includes a total of 5 questions for 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each question has 3 levels (no problems, some problems, and extreme problems). The EQ Visual Analogue Scale records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' (score of 100) and 'Worst imaginable health state' (score of 0).
Patients' quality of life, assessed by the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire. | at baseline and 12 months in the application group.(+18-and if applicable at 36 months/at the end of the study in the other intervention groups.) In the standard care groups at baseline and 12 or 18 months (and if applicable at the end of the study).
  The AFEQT is an atrial fibrillation-specific health-related quality of life questionnaire based on 18 questions in the domain of symptoms, daily activities and treatment concerns. A treatment satisfaction score can be calculated based on 2 additional questions. All questions are rated on a 7 point Likert scale. A scoring key is used to determine an overall AFEQT score and a treatment satisfaction score ranging from 0 to 100. A lower score indicates a worse health-related quality of life.
Patients' symptom burden, assessed by the Leuven ARrhythmia Questionnaire (LARQ). | at baseline,3- and 12 months in the application group.(+18-and if applicable at 36 months/at the end of the study in the other intervention groups).In the standard care groups at baseline and 12 or 18 months (and if applicable at the end of the study).
  The LARQ is based on 6 atrial fibrillation-related symptoms: palpitations, shortness of breath, chest pain, syncope, dizziness and fatigue. For each of these symptoms (except syncope), symptom prevalence, occurrence (frequency, duration, severity), distress, circumstances triggering the symptom, and effect on daily activities are requested. Subscale scores on five domains (symptom frequency, duration, effect on daily activities, severity and distress) are calculated by summing the raw scores and transforming them to a 0-100 scale. Higher scores represent a more pronounced symptom burden.
Patients' self-care capabilities, assessed by the Self-Care Questionnaire (SCQ). | at baseline, 3- and 12 months in the application group. (+18-and if applicable 36 months/at the end of the study in the other intervention groups).In the standard care groups at baseline and 12 or 18 months (and if applicable at the end of the study).
  This questionnaire includes a total of 15 questions. The first 6 questions will be scored on a 1 to 5 Likert scale. 1 is the best score and 5 is the worst score. The other 9 questions measure evolutions of self-care capabilities over time.
Patients' satisfaction of the intervention will be assessed by a study specific Patient Reported Outcome Measure (PROM) questionnaire. | at 12 months in all intervention groups and 12 or 18 months in the standard care groups.
  The number of questions will depend on the specific group allocation, ranging from a minimum of 4 questions to a maximum of 20 questions. These questions assess patients' satisfaction and opinion about the education provided during the study.

OTHER OUTCOMES:
The first occurrence of a cardiovascular event | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
  The first occurrence of a composite of cardiovascular death, a first cardiovascular hospitalization (i.e. hospitalization with overnight stay) and a first unplanned cardiovascular or neurological visit.
Mortality | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
  The occurrence of death will be followed.
Number of (un)planned hospital admissions | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
Hospital duration | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
Number of (un)planned cardiovascular and neurological visits | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
Number of cardiovascular emergency department visits | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
General practitioner visits | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
Exact time investments (in minutes) | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
  Time investments will be tracked (e.g. timing of the initiation session, the education sessions, feedback during medication telemonitoring, time spended on the application time and content usage).
Cost-utility analysis | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
  In all groups, the economic impact of hospitalizations, consultations, emergency department visits will be calculated using all relevant costs of inpatient and outpatient diagnostic/interventional procedures, based on the mean of hospital bills of each participating hospital. Since quality of life is evaluated throughout the trial, a cost-utility analysis will be performed.
Cost-effectiveness analysis | Patients (AF-EduCare study and AF-EduApp substudy) will be followed for a minimum of 12 months to a maximum of 36 months.
  In all groups, the economic impact of hospitalizations, consultations, emergency department visits will be calculated using all relevant costs of inpatient and outpatient diagnostic/interventional procedures, based on the mean of hospital bills of each participating hospital. With this data, a cost-effectiveness analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, MD, Phd, Principal Investigator — University Hospital of Antwerp
Locations (2):
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - Jessa Hospital, Hasselt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knaepen L, Desteghe L, Delesie M, Onder R, Vijgen J, Dendale P, Ector J, Heidbuchel H. Effectiveness of the AF-EduCare and AF-EduApp approach to improve atrial fibrillation knowledge and risk factor awareness in patients with atrial fibrillation: a randomized controlled trial. Eur J Cardiovasc Nurs. 2025 Mar 3;24(2):266-276. doi: 10.1093/eurjcn/zvae164. PMID 39780354
- [Derived] Delesie M, Knaepen L, Dendale P, Vijgen J, Ector J, Desteghe L, Heidbuchel H. Baseline demographics of a contemporary Belgian atrial fibrillation cohort included in a large randomised clinical trial on targeted education and integrated care (AF-EduCare/AF-EduApp study). Front Cardiovasc Med. 2023 Jun 2;10:1186453. doi: 10.3389/fcvm.2023.1186453. eCollection 2023. PMID 37332586